CLINICAL TRIAL: NCT00001339
Title: A Study of Combination Chemotherapy and Surgical Resection in the Treatment of Adrenocortical Carcinoma: Continuous Infusion Doxorubicin, Vincristine and Etoposide With Daily Mitotane Before and After Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930200; 93-C-0200
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-08

CONDITIONS: Adrenal Cortical Carcinoma
Keywords: Multidrug Resistance; Reversal of Drug Resistance; P-Glycoprotein; MDR-1
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Doxorubicin; Vincristine; Etoposide; Mitotane

INTERVENTIONS:
Drug: doxorubicin, vincristine, and etoposide with mitotane

SUMMARY:
Patients who have no response to preoperative chemotherapy and no residual disease following surgery on Regimen A are treated on Regimen B postoperatively.

The following acronyms are used:

DDD Mitotane, NSC-38721

DOX Doxorubicin, NSC-123127

VCR Vincristine, NSC-67574

VP-16 Etoposide, NSC-141540

Regimen A: 4-Drug Combination Chemotherapy followed by Surgery followed by 4-Drug Combination Chemotherapy. DDD/DOX/VCR/VP-16; followed by surgical debulking; followed by DDD/DOX/VCR/VP-16.

Regimen B: Single-Agent Chemotherapy. DDD.

DETAILED DESCRIPTION:
This is a study of infusional doxorubicin, vincristine, and etoposide in combination with daily oral mitotane in patients with adrenocortical cancer. Although mitotane has been used extensively in adrenocortical cancer and has documented single agent activity, only limited experience is available in the use of mitotane in combination with chemotherapy. In this trial the primary reason for using mitotane is an attempt to enhance therapeutic efficacy, based on its documented in-vitro activity as an antagonist of P-glycoprotein. The goal of this study is to determine the efficacy of this therapy by treating patients who are considered candidates for surgical resection at presentation or following a response to therapy. Following chemotherapy, patients deemed surgical candidates can undergo surgical resection with evaluation of response. Patients responding to chemotherapy will resume the combination treatment after surgery. Patients who do not respond will be maintained on single agent mitotane until it is deemed ineffective.

ELIGIBILITY:
Biopsy-proven primary or recurrent adrenocortical carcinoma considered surgically resectable at presentation or potentially resectable following an initial response to chemotherapy.

Potentially resectable disease includes primary lesion, nodal metastases, and liver and lung metastases if limited in size and number.

Patients for whom surgical resection is considered unlikely may be entered at the discretion of the investigator.

Measurable disease at presentation required.

A life expectancy of at least 3 months and a performance status (Karnofsky scale) of 70 percent or greater.

Prior chemotherapy is allowed, however, the patient should not have received chemotherapy four weeks before presentation.

Patients who have received prior doxorubicin may be enrolled provided they meet all other entry criteria and have an ejection fraction greater than 40 percent determined by MUGA scan.

Prior mitotane therapy is allowed. A dose of 3 gm/day should have been tolerated for at least one week. Patients do not need to be off mitotane therapy prior to starting this protocol.

WBC greater 3,000/mm(3); Platelet count greater than 100,000/mm(3); Creatinine clearance greater than 50 ml/min; bilirubin less than 1.5 mg/dl; serum transaminase less than 2 times normal.

Patient should be a good surgical candidate.

Must sign an informed consent and be geographically accessible to return for follow up treatment.

No presence of a second malignancy, other than squamous cell carcinoma of the skin.

No active systemic infection.

Must not be currently receiving treatment which cannot be discontinued with the following agents: diltiazem, nicardipine, phenothiazines, phenytoin, terfenadine or verapamil.

No positive serology for HIV.

No positive pregnancy test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42
Dates: Start 1993-08; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Luton JP, Cerdas S, Billaud L, Thomas G, Guilhaume B, Bertagna X, Laudat MH, Louvel A, Chapuis Y, Blondeau P, et al. Clinical features of adrenocortical carcinoma, prognostic factors, and the effect of mitotane therapy. N Engl J Med. 1990 Apr 26;322(17):1195-201. doi: 10.1056/NEJM199004263221705. PMID 2325710
- [Background] Bates SE, Shieh CY, Mickley LA, Dichek HL, Gazdar A, Loriaux DL, Fojo AT. Mitotane enhances cytotoxicity of chemotherapy in cell lines expressing a multidrug resistance gene (mdr-1/P-glycoprotein) which is also expressed by adrenocortical carcinomas. J Clin Endocrinol Metab. 1991 Jul;73(1):18-29. doi: 10.1210/jcem-73-1-18. PMID 1675220
- [Background] Cohn K, Gottesman L, Brennan M. Adrenocortical carcinoma. Surgery. 1986 Dec;100(6):1170-7. PMID 3787475